CLINICAL TRIAL: NCT06810960
Title: A 6-Year Postmarketing Safety and Clinical Outcome Study of Lecanemab in the Treatment of Alzheimer's Disease Using Real-World Data From South Korean Patients Enrolled Into the South Korean JOint RegistrY for ALZheimer's Treatment and Diagnostics (JOY-ALZ) Registry
Brief Title: A Postmarketing Study of Lecanemab in South Korean Participants With Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: BAN2401-M082-503
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Lecanemab; ARIA
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lecanemab: Participants treated with lecanemab in accordance with the approved prescribing information by a physician in routine clinical practice (postmarketing). Data will be collected from by JOY-ALZ registry.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The primary purpose of this study is to evaluate safety of lecanemab in the real-world clinical setting as reported by events of amyloid-related imaging abnormalities (ARIA)-edema (ARIA-E), ARIA-hemosiderin deposition (ARIA-H), symptomatic ARIA-E, symptomatic ARIA-H, and intracerebral hemorrhage (ICH) greater-than 1 centimeter (cm) in participants treated with lecanemab.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at consent
* Prior to JOY-ALZ enrollment, the treating physician confirms that the participant is suitable for lecanemab treatment, as per the approved indications in South Korea
* Has an identified study partner who provides separate written informed consent
* Provides written informed consent for the use of medical information to be shared with Eisai Korea Inc.

Exclusion Criteria:

* Currently participating in an interventional clinical study
* Has contraindications for lecanemab according to the approved prescribing information in South Korea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants prescribed with lecanemab by a physician in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events of Special Interest (AESIs) | Up to 6 years
  AESI will include ARIA-E, ARIA-H, symptomatic ARIA-E, symptomatic ARIA-H, and ICH greater-than 1 cm.
Exposure-adjusted Incidence Rate of AESIs | Up to 6 years
  AESI will include ARIA-E, ARIA-H, symptomatic ARIA-E, symptomatic ARIA-H, and ICH greater-than 1 cm.

SECONDARY OUTCOMES:
Incidence of Seizure, Anaphylaxis and Death | Up to 6 years
Exposure-Adjusted Incidence Rate of Seizure, Anaphylaxis and Death | Up to 6 years
Incidence of AESIs Based on Baseline Characteristics | Up to 6 years
  Baseline characteristics will include apolipoprotein E4 (APOE4) genotype, baseline magnetic resonance imaging (MRI) findings, prior Alzheimer's disease (AD) treatments, and antithrombotic therapy.
Exposure-adjusted Incidence Rate of AESIs Based on Baseline Characteristics | Up to 6 years
  Baseline characteristics will include APOE4 genotype, baseline MRI findings, prior AD treatments, and antithrombotic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai Trial Site #1, Nutley, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.